CLINICAL TRIAL: NCT06355739
Title: Phase II Clinical Study on the Safety and Efficacy of Autotransfusion Agents Targeting CD19 Chimeric Antigen Receptor T Lymphocytes (BIC-19GG, BIC-2019,BIC-2219)in the Treatment of CD19-positive Children With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma
Brief Title: CD19-targeted CAR T Cell Autotransfusion for the Treatment of Recurrent/Refractory B-cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma in Children With CD19+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhu Xiaofan (Other)
Responsible Party: Sponsor-Investigator, Zhu Xiaofan, Head of department, Institute of Hematology & Blood Diseases Hospital, China
Organization: Institute of Hematology & Blood Diseases Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIC-19GG, BIC-2019,BIC-2219
Record Dates: First submitted 2024-02-02; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: B Lymphocytic Leukemia; B Lymphoblastic Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 autotransfusion for B-cell acute lymphoblastic leukemia in children (Other)
  Interventions: Device: CAR T cell injection

INTERVENTIONS:
Device: CAR T cell injection — intravenous injection

SUMMARY:
To evaluate the safety and efficacy of BIC-19GG, BIC-2019, BIC-2219 in the treatment of relapsed/refractory B acute lymphoblastic leukemia/lymphoblastic lymphoma in children

ELIGIBILITY:
Inclusion Criteria:

1, age 3-18 years old (including boundary value), male and female;

2. The patient was clinically diagnosed as relapsed/refractory B acute lymphoblastic leukemia/lymphoblastic lymphoblastic

Patients with tumors who meet one of the following conditions:

• Complete marrow response (MRD>1%) or not achieved after at least 2 courses of standardized induction regimen chemotherapy

Complete response at the molecular level and immunology (characterized by specific molecular markers and immunophenotypes prior to treatment)

Patients, did not turn negative after treatment);

* Recurrence during chemotherapy, early recurrence after drug withdrawal (<12 months) or late recurrence after complete remission (≥

  12 months) and did not achieve complete remission after 1 course of standard induction regimen (MRD>1%);
* Recurrence after bone marrow transplantation;
* Simple bone marrow, simple extramedullary (testicular leukemia, central nervous system leukemia) or combined

recrudescence

3. Lansky score ≥60;

4, the treatment related antigen test result is positive (CD19/CD20/CD22);

5. The expected survival period from the signing date of the informed consent is more than 3 months;

6, HGB≥70g/L (blood transfusion);

7, liver and kidney function, cardiopulmonary function meet the following requirements:

1. Creatinine ≤1.5×ULN;
2. Left ventricular ejection fraction ≥50%;
3. Blood oxygen saturation >90%;
4. Total bilirubin ≤1.5×ULN; ALT and AST≤2.5 x ULN.-

   Exclusion Criteria:
   * 1, severe cardiac insufficiency, left ventricular ejection fraction <50%;

     2, have a history of severe lung function impairment;

     3. Combined with other advanced malignant tumors;

     4, combined with serious infection and can not be effectively controlled;

     5, combined with serious autoimmune disease or congenital immune deficiency;

     6, active hepatitis (hepatitis B virus deoxyribonucleic acid [HBVDNA] or hepatitis C virus ribonucleic acid [HCVRNA] positive);

     7, human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), or syphilis infection;

     8. Have a history of severe allergy to biological products (including antibiotics);

     9. Patients with allogeneic hematopoietic stem cell transplantation still had acute graft-versus-host response (GvHD) one month after immunosuppressant discontinuation;

     10, the presence of other serious physical or mental illnesses or abnormalities in laboratory tests that may increase the risk of participating in the study or interfere with the study results, as well as patients deemed unsuitable for participation in the study by the investigator.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival and event-free survival | 24 months post CAR-T cell infusion
  The prognosis of ALL children who underwent CAR-T cell therapy

SECONDARY OUTCOMES:
Overall remission rate | One month post CAR-T cell infusion
  The ORR of ALL children who underwent CAR-T cell therapy
Adverse events | 12 months post CAR-T cell infusion
  Incidence of adverse events and its severity

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Pediatrics, Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - InstituteHBDH, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No